CLINICAL TRIAL: NCT06259695
Title: Development and Usability of an Adjustable Prosthesis for Aquatic Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Laura Miller, Team Scientist II, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00219525
Record Dates: First submitted 2024-01-30; First posted 2024-02-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Amputation
Keywords: Aquatic Therapy; Limb Loss; Limb Difference; Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adjustable Aquatic Therapy Prosthesis (Experimental): The prosthesis will be designed to be adjustable in circumference, residual limb length, and overall height. This will allow adjustability to accommodate most limb shapes. The design will also provide secure suspension, on both land and in the water. This will maximize safety for the patient and translate motion from the residual limb to the prosthesis. Additionally, the prosthesis design will include a comfortable fit and interface, protecting the participant's skin. Skin will be assessed prior to use, during initial fitting, and after each therapy session. Finally, the prosthesis will be test fit and used with maximum assistance from clinical staff, minimizing risk.
  Interventions: Device: Adjustable Aquatic Therapy Prosthesis

INTERVENTIONS:
Device: Adjustable Aquatic Therapy Prosthesis — We will recruit up to three participants, who will attend up to two fitting appointments lasting up to one hour to assist in the design development. After the design of the prosthesis is completed, participants will attend three, 30-minute, aquatic therapy sessions with a physical therapist trained in aquatic therapy and utilize the prosthesis.

SUMMARY:
The initial purpose of this study is to develop a prosthesis which is adjustable to use with a variety of patients in aquatic therapy. Aquatic therapy is a beneficial rehabilitation tool for individuals with limb loss. The pool environment offloads body weight, which can improve comfort on a residual limb and increase confidence in activities outside of the pool. The properties of water also assist in strengthening exercises and reducing pain.

Currently, most individuals do not have a prosthesis to use in the pool. Water specific prosthesis are often not covered by insurance and can be expensive. For someone that doesn't have a water specific prosthesis, they may not be able to do therapy tasks on two legs, limiting what activities or exercises can be performed. Through creating an adjustable prosthesis, it will allow persons with limb loss to have access to a water specific leg in a time efficient, cost effective, and safe manner for rehabilitation.

This study involves a novel prosthesis for use in aquatic therapy. This novel design will have an adjustable circumference, residual limb length, and height, allowing a greater number of patients to use the prosthesis.

DETAILED DESCRIPTION:
The goal of this project is to create and conduct a preliminary usability evaluation of a novel adjustable prosthesis for use in aquatic therapy for persons with a lower limb amputation at the transtibial level (LLTTA). It is hypothesized that this prosthesis will benefit both the patient and the therapist during aquatic therapy sessions, which will be evaluated through the following aims:

Aim 1: Create a non-custom, adjustable prosthesis for use in aquatic therapy by individuals with limb loss at the transtibial level.

Aim 2: Perform a pilot study (n=3) to quantity the usability of the prosthesis as a therapy tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-89 years
* Patients who have a unilateral transtibial amputation who are able to use a prosthesis
* Patients who currently participate in aquatic therapy at Shirley Ryan AbilityLab, or have completed aquatic therapy within the last six months, at Shirley Ryan AbilityLab

Exclusion Criteria:

* Pregnant women
* Children (<18 years old)
* Prisoners or institutionalized individuals
* Individuals who have the inability to give informed consent
* Participants with complicating health conditions that interfere with the study
* Participants with contraindications to aquatic therapy, as listed in Shirley Ryan AbilityLab's policy on aquatic therapy participation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Survey - Subject | Through study completion, an average of one year.
  The System Usability Survey is a reliable tool for measuring the usability of a device. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.

SECONDARY OUTCOMES:
Socket Comfort Score | Through study completion, an average of one year.
  Rating system to assess prosthesis socket comfort. Scale ranges from 0-10, with 0 being the least comfortable and 10 the most comfortable.
System Usability Survey - Physical Therapist | Through study completion, an average of one year.
  The System Usability Survey is a reliable tool for measuring the usability of a device. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan Ability Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No